CLINICAL TRIAL: NCT02916264
Title: The Effect of Scalp Block on Surgical Pleth Index(SPI) During a Mayfield Head-holder Insertion in Neurosurgery : a Randomized Control Trial
Brief Title: The Effect of Scalp Block on Surgical Pleth Index(SPI) During a Mayfield Head-holder Insertion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Sirivimol Punjasawadwong, Principal Investigator, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03457
Record Dates: First submitted 2016-09-25; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Pain
Keywords: scalp block, surgical peth index
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a scalp block (Active Comparator): A standard scalp block ,with 0.5% bupivacaine total dose < 3 mg/kg, is performed by an anesthesiologist.
  Interventions: Procedure: a scalp block
- no scalp block (No Intervention): An anesthesiology will pretend to perform the scalp block,

INTERVENTIONS:
Procedure: a scalp block — Bilateral blocks of six nerves: ie. supraorbital and supraorbital nerves (V1), zygomaticotemporal nerves (V2) , auriculotemporal nerves , greater occipital nerves, and lesser occipital nerves will be performed by a well trained anesthesiologist with 0.5% bupivacaine not exceeding 3 mg/kg
  Arms: a scalp block

SUMMARY:
It is a randomized control trial to compare the surgical plethysmographic index (SPI) response during a Mayfield head-holder insertion in neurosurgical patients who receive a scalp block versus those who do not receive the scalp block after induction of anesthesia with propofol with fentanyl and intubation with cis-atracurium.

DETAILED DESCRIPTION:
Study design is a randomized controlled trial Participants include adult neurosurgical patients scheduled to have a Mayfield head-holder insertion for supratentorial craniotomy Intervention is a scalp block prior to a Mayfield head holder insertion. Comparison is 'no scalp block' Outcome is surgical plethysmographic index (SPI) responses during/after a Mayfield head holder insertion Sample size includes 30 cases (15 cases per arm)

The eligible neurosurgical patients will be randomly allocated, by a concealed randomization process, to receive or not to receive a scalp block after induction and intubation with propofol/fentanyl and cisatracurium. Surgical plethysmographic index, direct arterial blood pressure, heart rate (EEG), End tidal Carbondioxide, Bispectral/entropy (40-60) will be recorded every one minute before/after induction and intubation, before/after the scalp block, and before/after the Mayfield head-holder insertion. The Mayfield head-holder insertion will be performed by a neurosurgeon who will be blinded to the allocated groups.

Data analysis is performed to compare the change of SPI during and after the Mayfield head-holder insertion from the baseline in both groups by using repeated measure ANOVA at the significant level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients will receive a Mayfield head-holder insertion for supratentorial craniotomy

Exclusion Criteria:

* History of chronic hypertension, Diabetes mellitus (DM), coronary heart diseases
* Receiving beta blockers
* BMI > 30
* Coagulopathy
* severe liver and renal diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
the change of SPI from baseline | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sirivimol Punjasawadwong, MD, Principal Investigator — Dpt Anesthesiology, Faculty of Medicine, Chiang Mai University
Locations (1):
- Dpt Anesthesiology, Faculty of Medicine, Chiang Mai University, Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided